CLINICAL TRIAL: NCT06787612
Title: Multi-arm Phase 2 Study of Ubamatamab (REGN4018; MUC16×CD3 Bispecific Antibody) With or Without Additional Agents in Platinum-Resistant Ovarian Cancer
Brief Title: Investigation of Ubamatamab Combination Therapy in Adult Participants With Platinum-Resistant Ovarian Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R4018-ONC-2445; 2024-517806-27-00 (Registry Identifier: EUCT Number)
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-10

CONDITIONS: Ovarian Cancer
Keywords: Platinum Resistance; Fallopian Tube Cancer; Primary Peritoneal Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Bevacizumab; cemiplimab; 1-dodecylpyridoxal; liposomal doxorubicin; sarilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm A1 (Experimental): Randomization as described in the protocol
  Interventions: Drug: Ubamatamab; Drug: Sarilumab
- Arm A2 (Experimental): Randomization as described in the protocol
  Interventions: Drug: Ubamatamab; Drug: Sarilumab
- Arm B (Experimental): Randomization as described in the protocol
  Interventions: Drug: Ubamatamab; Drug: Bevacizumab; Drug: Sarilumab
- Arm C (Experimental): Randomization as described in the protocol
  Interventions: Drug: Ubamatamab; Drug: Cemiplimab; Drug: Fianlimab; Drug: Sarilumab
- Arm D (Experimental): Randomization as described in the protocol
  Interventions: Drug: Ubamatamab; Drug: PLD; Drug: Sarilumab

INTERVENTIONS:
Drug: Ubamatamab — Administered per the protocol
  Other Names: REGN4018
Drug: Bevacizumab — Administered per the protocol
  Other Names: Avastin®
  Arms: Arm B
Drug: Cemiplimab — Administered per the protocol
  Other Names: Libtayo®; REGN2810
  Arms: Arm C
Drug: Fianlimab — Administered per the protocol
  Other Names: REGN3767
  Arms: Arm C
Drug: PLD — Administered per the protocol
  Other Names: Doxil®; Pegylated liposomal doxorubicin
  Arms: Arm D
Drug: Sarilumab — Prophylaxis administered per the protocol
  Other Names: Kevzara®; REGN88; SAR153191

SUMMARY:
This study is researching an experimental drug called ubamatamab, also referred to as "study drug". The study is focused on patients who have advanced ovarian cancer.

The aim of the study is to see how safe, tolerable, and effective the study drug is on its own and in combination with other anti-cancer drugs (bevacizumab, cemiplimab, fianlimab and a standard chemotherapy drug, pegylated liposomal doxorubicin [PLD]), referred to as "combination drugs'.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drug and its experimental combinations
* How much study drug and fianlimab is in the blood at different times
* Whether the body makes antibodies against the study drug (which could make the drug less effective or could lead to side effects) and its combinations

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants with histologically or cytologically confirmed diagnosis of advanced serous or endometrioid ovarian, primary peritoneal, or fallopian tube cancer (clear cell, mucinous, and carcinosarcoma are excluded)
2. Must have progression on prior therapy documented radiographically and must have at least 1 measurable lesion (not previously irradiated) that can be accurately measured by RECIST 1.1
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Adequate organ and bone marrow function, as described in the protocol
5. Platinum-Resistant Ovarian Cancer, as described in the protocol

Key Exclusion Criteria:

1. Major surgical procedure or significant traumatic injury within 4 weeks prior to first dose of study drug(s)
2. Documented allergic or acute hypersensitivity reaction attributed to antibody treatments or doxorubicin hydrochloride or components of study drug(s)
3. Another malignancy that is progressing or requires active treatment, as described in the protocol
4. Untreated or active primary brain tumor, Central Nervous System (CNS) metastases, or spinal cord compression, as described in the protocol
5. Uncontrolled infections including but not limited to human immunodeficiency virus, hepatitis B or hepatitis C infection, or diagnosis of immunodeficiency

NOTE: Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 220 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2028-12-07 (Estimated); Study Completion 2028-12-07 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 by investigator assessment | Up to 3 years

SECONDARY OUTCOMES:
Cancer Antigen (CA) -125 response by Gynecologic Cancer Intergroup (GCIG) Criteria | Up to 3 years
Complete Response (CR) rate by RECIST 1.1 | Up to 3 years
Disease Control Rate (DCR) by RECIST 1.1 | Up to 3 years
Duration Of Response (DOR) by RECIST 1.1 | Up to 3 years
Progression-Free Survival (PFS) by RECIST 1.1 | Up to 3 years
Incidence of Grade ≥ 2 Cytokine Release Syndrome (CRS) by Lee criteria | Up to 3 years
Treatment-Emergent Adverse Events (TEAEs) by Common Terminology Criteria for Adverse Events (CTCAE) v5.0 | Up to 3 years
TEAEs by Lee criteria | Up to 3 years
Concentration of ubamatamab in serum over time | Up to 3 years
Concentration of fianlimab in serum over time | Up to 3 years
Incidence of anti-drug antibodies (ADA) to ubamatamab | Up to 3 years
Titer of ADA to ubamatamab | Up to 3 years
Incidence of ADA to fianlimab | Up to 3 years
Titer of ADA to fianlimab | Up to 3 years
Incidence of ADA to cemiplimab | Up to 3 years
Titer of ADA to cemiplimab | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (43):
- United States (16):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - UC San Diego Health, La Jolla, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Tampa General Hospital Cancer Institute, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Norton Cancer Institute, St. Matthews Clinic, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - The Ohio State University Comprehensive Cancer Center, Hilliard, Ohio
  - Providence Cancer Institute, Portland, Oregon
  - Avera Cancer Institute Sioux Falls, Sioux Falls, South Dakota
  - Swedish Cancer Institute, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- South Korea (10):
  - National Cancer Center, Gyeonggi-do, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon, Seoul
  - Keimyung University Dongsan Hospital, Daegu
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Univ. of Ulsan, Seoul
  - Samsung Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Korea University Guro Hospital, Seoul
- Taiwan (7):
  - Changhua Christian Hospital, Changhua, Changhua City
  - Chi Mei Medical Center, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Taipei Municipal Wan Fang Hospital, Taipei
- Turkey (Türkiye) (10):
  - Medicalpark Seyhan Hospital, Seyhan, Adana
  - Hacettepe University, Altındağ, Ankara
  - Medipol University Hospital, Istanbul, Bagcilar
  - Gaziantep Medicalpoint Hospital, Gaziantep, Sehitkamil
  - Baskent University, Adana
  - Sbu Doctor Abdurrahman Yurtaslan Ankara Onkoloji Suam, Ankara
  - Ankara Bilkent City Hospital, Ankara
  - Memorial Ankara Hospital, Ankara
  - Cerrahpasa Medical Faculty At Istanbul University Cerrahpasa, Istanbul
  - Sakarya University - Education and Research Hospital, Sakarya

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/